CLINICAL TRIAL: NCT03390530
Title: Thyroxine Treatment in Premature Infants With Intraventricular Hemorrhage: Phase III Clinical Trial
Brief Title: Thyroxine Treatment in Premature Infants With Intraventricular Hemorrhage
Acronym: IVHT4
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed by PI prior to approval
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Westchester Medical Center (Other); Morgan Stanley Children's Hospital (Other); University of Pittsburgh (Other); Children's Minnesota Hospital (Unknown); University of Minnesota (Other); St. Louis University (Other); Arkansas Children's Hospital Research Institute (Other); Brigham and Women's Hospital (Other); University of North Carolina, Chapel Hill (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Praveen Ballabh, Professor of Pediatrics, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-8707
Record Dates: First submitted 2017-12-21; First posted 2018-01-04 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Intraventricular Hemorrhage of Prematurity
Keywords: Thyroxine; Intraventricular hemorrhage; MRI with DTI,; Neurodevelopmental outcome
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: Double-blinded, placebo-controlled, and randomized controlled trial to compare outcomes between thyroxine and placebo treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded and randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Thyroxine treatment (Active Comparator): Intravenous thyroxine in a dose of 8 µg/kg/day divided into two doses (every 12 hours)
  Interventions: Drug: Thyroxine
- Placebo treatment (Placebo Comparator): Intravenous placebo treatment every 12 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thyroxine — 8 µg/kg/day divided into two doses intravenous every 12 hours
  Other Names: Levothyroxine
  Arms: Thyroxine treatment
Drug: Placebo — Placebo
  Other Names: Inactive substance in a similarly looking solution
  Arms: Placebo treatment

SUMMARY:
Brain bleed in premature infants damages the brain and survivors suffer from cerebral palsy (weakness in the extremities), cognitive deficits, and neurobehavioral disorders. In this clinical trial, investigators will test whether thyroxine (hormone from thyroid gland) treatment in premature infants with moderate-to-large brain bleeds show recovery in the brain structure on MRI evaluation at the time of discharge (44+/-1 weeks) and neurodevelopmental improvement at 2 years of age.

DETAILED DESCRIPTION:
Intraventricular hemorrhage (IVH) remains a major complication of prematurely born infants. Survivors of IVH suffer from cerebral palsy, cognitive deficits and neurobehavioral disorders. In the proposed study We hypothesize that T4 treatment in preterm (230/7-276/7 weeks) infants with grade II-IV IVH will: a) improve MRI biomarkers, including total myelinated white matter volume, Kidokoro scoring, functional connectivity between motor brain regions, and fractional anisotropy in the corpus callosum of preterm infants with grade II-IV IVH at 36 weeks postmenstrual age, and b) better composite outcome of disability and death. The composite outcome will be derived by integrating scores for Bayley Scales of Infant and Toddler Development (BSID-IV) Motor subscale at 22-26 months in survivors and BSID IV value of 46 assigned to deceased infants. To test these hypotheses, we will perform a randomized double-blinded placebo-controlled trial to determine the effect of T4 treatment on preterm infants with grade II-IV IVH. Ten participating neonatal intensive care units will enroll 346 premature infants (230/7-276/7 weeks gestational age. 173 in each arm) with unilateral or bilateral grade II-IV IVH over a period of 3 years. The treatment will consist of T4 administration (8 µg/kg/day divided into two doses) up to 34 weeks of postmenstrual age, which will be initiated at 2-5 days of postnatal age in all cases. The infants will undergo MRI with DTI at 36 weeks and neurobehavioral evaluation at 22-26 months of corrected age. We have assumed a 7.5 point mean difference (SD=15) in BSID-IV motor subscale between T4 and placebo groups, an overall mortality rate of 25%, and 5% reduction in mortality for each SD change in outcome. Based on these, we expect an increase in the induced composite outcome by ≥5.6 points in T4 treated group compared to placebo controls. The study will conclusively determine whether the proposed clinical trial of T4 treatment enhances motor outcome and diminishes composite endpoint of death or disability in preterm infants with grade II-IV IVH.

ELIGIBILITY:
Inclusion Criteria

* NICU inpatients born between 23-0/7 and 27-6/7 weeks of gestation
* Postnatal age 3-6days (≥3 d ≤ 6 d)
* Unilateral or bilateral Grade 3 or 4 IVH
* Parental consent

Exclusion criteria:

* Major malformations, including surgical, cardiac, cerebral, chromosomal, or genetic syndromes, identifiable at or before birth;
* Congenital bacterial infection proven by culture at birth or viral syndrome known prior to delivery (e.g. chicken pox, rubella, etc.)

Ages: 3 Days to 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-01-18 (Estimated); Primary Completion 2025-12-18 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
Death or disability | 22-26 months of age
  The primary outcome will be a quantitative composite outcome using the BSID-IV Motor score measured at 22-26 months among survivors while incorporating death using a floor value of 46.

SECONDARY OUTCOMES:
BSID-IV Motor subscale | 22-26 months of age
  Bayley Scales of Infant and Toddler Development (BSID) IV score.
BSID-IV Cognitive subscale | 22-26 months of age
  Bayley Scales of Infant and Toddler Development (BSID) IV score.
BSID-IV Language subscale | 22-26 months of age
  Bayley Scales of Infant and Toddler Development (BSID) IV score.
Binary composite outcome of death or moderate/severe NDI | 22-26 months of age
  NDI will be defined as the presence of any of the following: BSID-IV Cognitive < 85, BSID-IV Motor <85, GMFCS ≥ 2 (NICHD, Neonatal Res. Network 2018)
Cerebral palsy incidence and severity | 22-26 months of age
  We will perform neurological examination as in PENUT study and GMFCS scoring to determine cerebral palsy incidence and severity

OTHER OUTCOMES:
MRI studies: dMRI measures (fractional anisotropy; radial, axial and mean diffusivity) in the corpus callosum and corticospinal tract | 44+/-1 weeks of postmenstrual age
  dMRI analyses
MRI studies: myelinated and unmyelinated WM brain volume | 44+/-1 weeks of postmenstrual age
  After visual quality control, initial total brain segmentation for tissue types will be done using T2 weighted images with MANTIS, an in-house method of automated Morphologically Adaptive Neonatal Tissue Segmentation (Alexander, et al. 2017)
MRI studies: Kidokoro WM and global scores | 44+/-1 weeks of postmenstrual age
  Kidokoro WM and global scores as in Kidokoro et al ( Am J Neuroradiol 34, 2208-2214:2013)

CONTACTS AND LOCATIONS:
Overall Officials: PRAVEEN BALLABH, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Praveen Ballabh, The Bronx, New York, United States